CLINICAL TRIAL: NCT02616523
Title: Influence of Dexmedetomidine and Lidocaine on Opioid Consumption, Cognitive Function and Incidence of Neuropathic Pain in Laparoscopic Intestine Resection
Brief Title: Influence of Dexmedetomidine and Lidocaine on Opioid Consumption in Laparoscopic Intestine Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Lea Andjelkovic, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23/07/14
Record Dates: First submitted 2015-11-07; First posted 2015-11-30 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Opioid-Related Disorders; Neuralgia
Keywords: dexmedetomidine; lidocaine; neuropathic pain; laparoscopic intestine resection; cognitive function
MeSH Terms: conditions — Opioid-Related Disorders; Neuralgia | interventions — Dexmedetomidine; Lidocaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- dexmedetomidine (Active Comparator): The investigators will compare fentanyl consumption in participants undergoing laparoscopic intestine resection intra and postoperatively. Dexmedetomidine group will receive dexmedetomidine infusion 0,5 mcg/kg/h beside boluses of fentanyl.
  Interventions: Drug: Dexmedetomidine; Drug: Fentanyl
- lidocaine (Active Comparator): Lidocaine group will receive lidocaine infusion 1,5 mg/kg/h during the laparoscopic intestine resection.
  Interventions: Drug: Lidocaine; Drug: Fentanyl
- placebo (Placebo Comparator): The placebo group will receive intravenous infusion of normal saline only.
  Interventions: Other: placebo; Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — The participants will be given infusion of dexmedetomidine 0,5 mcg/kg/h intravenously.
  Other Names: Dexdor
  Arms: dexmedetomidine
Drug: Lidocaine — The participants will be given infusion of lidocaine 1,5 mg/kg/h intravenously.
  Other Names: Xylocaine
  Arms: lidocaine
Other: placebo — The participants will be given infusion of normal saline intravenously.
  Arms: placebo
Drug: Fentanyl — Fentanyl 2 mcg/kg will be given to all participants for the intubation and during the operation when ANI value drops below 50.

SUMMARY:
Using combination of opioid analgesics and analgesics with different mechanism of action the investigators can decrease the consumption of opioid analgesics and their side effects. The investigators will use opioid analgesic fentanyl alone or in combination with dexmedetomidine or lidocaine.The participants scheduled for laparoscopic intestine resection will be divided in three groups: in the first group, the participants will receive single boluses of fentanyl, in the second group, the participants will receive continuous infusion of lidocaine and single boluses of fentanyl, and in the third group, the participants will receive continuous infusion of dexmedetomidine and single boluses of fentanyl. Participants with intraoperative infusion od dexmedetomidine or lidocaine will need less boluses of fentanyl during the operation and less opioid analgesics after the operation in comparison to those who will receive only fentanyl boluses. Better cognitive function after the operation is expected in participants receiving dexmedetomidine infusion. There will be minimal incidence of neuropathic pain because of minimal surgical injury of peripheral nerves in all groups of patients.

DETAILED DESCRIPTION:
Introduction: The consumption of opioid analgetics and their side effects can be minimized by using the combination of opioid analgesics and analgesics with different mechanism of action. The investigators will use opioid analgesic fentanyl alone or in combination with dexmedetomidine or lidocaine. Dexmedetomidine is alpha 2 adrenergic receptor agonist and is used more and more during anesthesia because of its anesthetic and analgesic effects as it preserves mental status and decreases the consumption of analgesics. Lidocaine is a local anesthetic and antiarrhythmic drug which decreases opioid consumption as well.

The participants scheduled for laparoscopic intestine resection will be divided in three groups: in the first group, the participants will receive single boluses of fentanyl, in the second group, the participants will receive continuous infusion of lidocaine and single boluses of fentanyl, and in the third group, the participants will receive continuous infusion of dexmedetomidine and single boluses of fentanyl.

Hypothesis: Participants with intraoperative infusion od dexmedetomidine or lidocaine will need less boluses of fentanyl during the operation and less opioid analgesics after the operation in comparison to those who will receive only fentanyl boluses. Better cognitive function after the operation in participants receiving dexmedetomidine infusion is expected. There will be minimal incidence of neuropathic pain because of minimal surgical injury of peripheral nerves in all groups.

Justification: Lidocaine and dexmedetomidine are analgesics with different mechanism of action in comparison to opioid analgesics. Their use during the operation decreases the consumption of opioids intra- and postoperatively. Dexmedetomidine has beneficial effect on cognitive function and that is why the investigators expect preserved cognitive function in participants after the operation. Because of minimal surgical injury and, therefore, minimal probability of peripheral nerve injury, the investigators expect low incidence of neuropathic pain in all groups.

Methods: The investigators will include 60 participants in the study, between 35 to 85 years old, ASA 2 - 3 (American Society of Anesthesiologists, ASA) undergoing a planned laparoscopic intestine resection. The participants will be randomized into three groups. In the first group, fentanyl boluses will be adimistred during the operation, in the second, infusion of lidocaine will be added to fentanyl, and in the third, the infusion of dexmedetomidine will be added to fentanyl. The investigators will record opioid consumption during the operation and two days after the operation. The investigators will use mini mental test for evaluation of cognitive function before the operation and at the transfer of the participant postoperatively to the surgical ward, in order to explore the influence of analgesics used on cognitive function. Two months after the operation the degree of neuropathic pain will be evaluated with pain questionnaire. The data will be statistically evaluated.

Expected results: Participants with intraoperative infusion of lidocaine and dexmedetomidine will need less opioid analgesics during and after the operation in comparison to the group with fentanyl boluses only. The investigators expect better cognitive function after the operation in participants with dexmedetomidine infusion. Because of the minimal surgery injury to the peripheral nerves low incidence of neuropathic pain is expected in all groups.

Study design and methods Inclusion criteria: In our study the investigators will include patients aged 35 to 85, ASA 2-3 (according to the classification of American Society of Anesthesiologists), undergoing a planned laparoscopic intestine resection at the Department of Abdominal Surgery at the University Medical Centre Ljubljana. Included participants will sign the consensus for participating in the study after exact explanation and conversation, as well as consensus for anesthesia and surgery.

Exclusion criteria: Participants with allergies to alpha 2 receptor agonists, uncontrolled arterial hypertension, 2nd and 3rd degree atrioventricular block, alcohol and illegal drugs abusers, patients with clinically important neurological, cardiovascular, respiratory (COPD, emphysema), renal, liver, and gastrointestinal disease, will be excluded from our study. The investigators will also exclude pregnant women and patients younger than 18 years due to their physiological particularities.

Data collection: The participants will be prepared for the operation as usual according to the operative protocol. Cognitive function is going to be assessed with a mini mental test before the operation.

After inserting the peripheral venous line, the induction will be performed with analgesic fentanyl (2 mcg/kg) and sedative propofol (1,5-2,5 mg/kg). Muscle relaxant rocuronium will be used for easier intubation (0,6 mg/kg; standard dose). The participants will be controlled mechanically ventilated with tidal volumes 6-8 ml/kg. Anesthesia will be maintained with intravenous anesthetic propofol in doses between 4 - 6 mg/kg/h according to bispectral index value (bispectral index, BIS, Vista), which will be kept between 40 and 55, the interval suitable for surgical depth of anesthesia. Normothermia and normocapnia will be maintained. The fluids will be warmed to 39°C via Hotline, the body temperature and expired CO2 will be measured. Mean arterial blood pressure will be maintained within ± 25 % baseline value. When mean arterial blood pressure will decrease more than 25% from the baseline value, a bolus of a vasoactive drug will be used.

Beside the standard monitoring (electrocardiogram, pulse oximetry, indirect blood pressure management, capnometry), the investigators will use ANI (analgesia nociception index) monitoring for the pain measurement. ANI values will be maintained between 50 and 70 and between those valuse good analgesia is provided. Muscle relaxation will be measured with TOF (train of four) and will be maintained on the level of deep muscle relaxation, that is TOF 0 and PTC 1 - 2 (posttetanic count).

Before the operation the investigators will randomize the participants into the three groups, which will distinguish according to analgesia used. All participants will get intravenous bolus of fentanyl (2 mcg/kg, standard dose) before the incision. All of them will receive bolus of fentanyl when ANI will drop below 50 during the operation (2 mcg/kg, recommended standard dose, first group). Participants in the second group will receive infusion of lidocaine (1,5 mg/kg/h), and participants in the third group infusion of dexmedetomidine (0,5 µg/kg/h). The consumption of fentanyl and propofol will be measured during the operation. The infusion of lidocaine and dexmedetomidine will be stopped 10 minutes before the end of the operation. Propofol infusion will be stopped at the end of the final suture. After the operation all participants will receive postoperative infusion of piritramide delivered with PCA (patient control analgesia). If the pain according to the visual analog scale (VAS) will be more than 3, the participants will be given a bolus of the peripheral acting analgesic or opioid (paracetamol, metamizol, piritramide). VAS will be reevaluated two days after the operation, as well as the consumption of other opioids and other analgesics. Cognitive function will be evaluated again on the second day with mini mental test, or at the transfer of the participant to the surgical ward with the discontinuation of the opioids and when they will be afebrile. Neuropathic pain will be evaluated with the pain questionnaire two months after the operation.

Statistical analysis: Collected data will be presented using descriptive statistics such as mean, median and standard deviation. The use of the opioids and other analgesics will be compared using paired Student t-test or other suitable nonparametric tests (eg. ANOVA), depending on the type of data used.

Correlation of different factors will be determined using Pearson/Spearman correlation coefficient. Deviation from normal distribution of data will be tested with a chi-squared test. Predictive value will be determined using logistic regression.

Expected results: The investigators assume that there will be less opioid consumption in participants receiving lidocaine or dexmedetomidine infusion during the operation and the following two days compared to participants who received fentanyl boluses only. In participants with intraoperative infusion of dexmedetomidine the investigators expect preserved cognitive function. Low incidence of neuropathic pain is expected two months after the operation in all groups because of minimal peripheral nerve injury during operation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 35 to 85,
* ASA 2-3 (according to the classification of American Society of Anesthesiologists),
* undergoing a planned laparoscopic intestine resection at the Department of Abdominal Surgery at the University Medical Centre Ljubljana.

Exclusion Criteria:

* allergies to alpha 2 receptor agonists,
* uncontrolled arterial hypertension,
* 2nd and 3rd degree atrioventricular block,
* alcohol and illegal drugs abusers,
* patients with clinically important neurological, cardiovascular, respiratory (COPD, emphysema), renal, liver, and gastrointestinal disease,
* pregnant women,
* patients younger than 18 years-

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lea Andjelkovic, MD, Principal Investigator — UMC Ljubljana Slovenia

REFERENCES:
- [Background] Vigneault L, Turgeon AF, Cote D, Lauzier F, Zarychanski R, Moore L, McIntyre LA, Nicole PC, Fergusson DA. Perioperative intravenous lidocaine infusion for postoperative pain control: a meta-analysis of randomized controlled trials. Can J Anaesth. 2011 Jan;58(1):22-37. doi: 10.1007/s12630-010-9407-0. PMID 21061107
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Background] Tufanogullari B, White PF, Peixoto MP, Kianpour D, Lacour T, Griffin J, Skrivanek G, Macaluso A, Shah M, Provost DA. Dexmedetomidine infusion during laparoscopic bariatric surgery: the effect on recovery outcome variables. Anesth Analg. 2008 Jun;106(6):1741-8. doi: 10.1213/ane.0b013e318172c47c. PMID 18499604
- [Background] Shin JH, Howard FM. Abdominal wall nerve injury during laparoscopic gynecologic surgery: incidence, risk factors, and treatment outcomes. J Minim Invasive Gynecol. 2012 Jul-Aug;19(4):448-53. doi: 10.1016/j.jmig.2012.03.009. Epub 2012 May 3. PMID 22560041
- [Background] Niccolai P, Ouchchane L, Libier M, Beouche F, Belon M, Vedrinne JM, El Drayi B, Vallet L, Ruiz F, Biermann C, Duchene P, Chirat C, Soule-Sonneville S, Duale C, Dubray C, Schoeffler P. Persistent neuropathic pain after inguinal herniorrhaphy depending on the procedure (open mesh v. laparoscopy): a propensity-matched analysis. Can J Surg. 2015 Apr;58(2):114-20. doi: 10.1503/cjs.008314. PMID 25799247
- [Background] Spindler Vesel A, Vrečar V, Repar A, Požar Lukanović N. Efficiency of PCA with piritramid and postoperative occurence of neuropathic pain in laparoscopic and clasical colorectal surgery. In: Della Roca G, De Monte A, eds. Proceedings of 25th Anesthesia And ICU Symposium Alpe-Adria. Udine, 2012:90-3.
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Jeanne M, Logier R, De Jonckheere J, Tavernier B. Heart rate variability during total intravenous anesthesia: effects of nociception and analgesia. Auton Neurosci. 2009 May 11;147(1-2):91-6. doi: 10.1016/j.autneu.2009.01.005. Epub 2009 Feb 8. PMID 19201661
- [Background] Penney R. Use of dexmedetomidine and ketamine infusions during scoliosis repair surgery with somatosensory and motor-evoked potential monitoring: a case report. AANA J. 2010 Dec;78(6):446-50. PMID 21309291
- [Background] Feld JM, Hoffman WE, Stechert MM, Hoffman IW, Ananda RC. Fentanyl or dexmedetomidine combined with desflurane for bariatric surgery. J Clin Anesth. 2006 Feb;18(1):24-8. doi: 10.1016/j.jclinane.2005.05.009. PMID 16517328
- [Background] McCarthy GC, Megalla SA, Habib AS. Impact of intravenous lidocaine infusion on postoperative analgesia and recovery from surgery: a systematic review of randomized controlled trials. Drugs. 2010 Jun 18;70(9):1149-63. doi: 10.2165/10898560-000000000-00000. PMID 20518581
- [Derived] Andjelkovic L, Novak-Jankovic V, Pozar-Lukanovic N, Bosnic Z, Spindler-Vesel A. Influence of dexmedetomidine and lidocaine on perioperative opioid consumption in laparoscopic intestine resection: a randomized controlled clinical trial. J Int Med Res. 2018 Dec;46(12):5143-5154. doi: 10.1177/0300060518792456. Epub 2018 Sep 13. PMID 30209962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between June 2014 and April 2015 at Ljubljana University Medical Centre, Slovenia.
Pre-assignment Details: We excluded from the study: the participants with allergies to α2 receptor agonists, uncontrolled arterial hypertension, 2nd and 3rd degree atrioventricular block, alcohol abusers, clinically important neurological, cardiovascular, respiratory, renal, liver, and gastrointestinal disease, pregnant women and participants younger than 18 years.
Period: Overall Study
Arm/Group | Dexmedetomidine | Lidocaine | Placebo
Started | 20 (June 2014) | 20 (June 2014) | 20 (June 2014)
Completed | 19 (April 2015) | 20 (April 2015) | 20 (April 2015)
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexmedetomidine | Lidocaine | Placebo | Total
Number analyzed (Participants) | 19 | 20 | 20 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (12) | 61 (11) | 58 (12) | 62 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 10 | 28
  Male | 9 | 12 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Consumption of Fentanyl
Description: consumption of fentanyl (mg) during the procedure
Time Frame: time of the operation
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Dexmedetomidine | Lidocaine | Placebo
Number analyzed (Participants) | 19 | 20 | 20
mg | 41 (10) | 50 (18) | 58 (21)

2. Secondary Outcome: Consumption of Piritramide
Description: consumption of piritramide (mg) in the recovery room
Time Frame: one hour after the operation
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Dexmedetomidine: Participants received dexmedetomidine infusion intraoperatively 0,5 mcg/kg/h
- Lidocaine: Participants received lidocaine infusion intraoperatively 1,5 mg/kg/h
- Placebo: Participants received fentanyl boluses during the operation
Arm/Group | Dexmedetomidine | Lidocaine | Placebo
Number analyzed (Participants) | 19 | 20 | 20
mg | 4.63 (4.95) | 5.25 (7.04) | 4.25 (2.95)

3. Secondary Outcome: Neuropathic Pain (Pain Questionnaire) dn4
Description: Pain questionnaire dn4 will be send to participants after two months of surgery to evaluate the neuropathic pain. There are minimum 0 points and maximum 10 points. If the score is 4 or higher then the pain is likely to be neuropathic pain.
Time Frame: two months after the surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dexmedetomidine | Lidocaine | Placebo
Number analyzed (Participants) | 19 | 20 | 20
units on a scale | 0.11 (0.46) | 0.00 (0.00) | 0.45 (0.83)

4. Other Pre Specified Outcome: Complication
Description: complications such as obstipation in the postoperative period
Time Frame: up to two weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Dexmedetomidine | Lidocaine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Limitations of our study is that we have not evaluated inflammatory response on the cellular level. This should be investigated in the future studies to establish if dexmedetomidine and lidocaine have clinically important anti-inflammatory effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No